CLINICAL TRIAL: NCT00618059
Title: A Single Dose, Two-Period, Two-Treatment, 2-Sequence Crossover Bioequivalency Study of 7.5 mg Pilocarpine Tablets Under Fed Conditions
Brief Title: Bioequivalency Study of 7.5 mg Pilocarpine Under Fed Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roxane Laboratories (Industry)
Responsible Party: Elizabeth Ernst, Director, Drug Regulatory Affairs and Medical Affairs, Roxane Laboratories, Inc.
Organization: West-Ward Pharmaceutical (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PILO-04
Record Dates: First submitted 2008-01-15; First posted 2008-02-18 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Dry Mouth
MeSH Terms: conditions — Xerostomia | interventions — Pilocarpine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Pilocarpine

SUMMARY:
The objective of this study was the bioequivalence of a Roxane Laboratories' Pilocarpine tablets, 7.5 mg, to SALAGEN® Tablets, 7.5 mg (MGI) under fed conditions using a single-dose, randomized, 2-treatment, 2-period, 2-sequence crossover design.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal findings on the physical examination, medical history, or clinical laboratory results during screening.

Exclusion Criteria:

* Positive test for HIV, Hepatitis B, or Hepatitis C.
* Treatment with known enzyme altering drugs.
* History of allergic or adverse response to Pilocarpine or any comparable or similar product.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2004-08; Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Bioequivalence | Baseline, Two period, Seven day washout

CONTACTS AND LOCATIONS:
Overall Officials: Daniel V Freeland, DO, Principal Investigator — CEDRA Clinical Research, LLC
Locations (1):
- CEDRA Clinical Research, LLC, Austin, Texas, United States